CLINICAL TRIAL: NCT05166460
Title: Novel Cooling Device for the Elimination of Warm Ischemia During Renal Transplantation
Acronym: QuitWIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Thomas Skinner (Other)
Collaborators: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor-Investigator, Thomas Skinner, Principal Investigator, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Device Feasibility
Other Study IDs: 1026704
Record Dates: First submitted 2021-07-06; First posted 2021-12-22 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Kidney Transplant; Complications; Delayed Graft Function
Keywords: kidney; transplant; warm ischemia time; delayed graft function; vascular anastomosis; renal hypothermia
MeSH Terms: conditions — Delayed Graft Function

STUDY DESIGN:
Intervention Model Description: 1:1 randomization (Part B, 40 patients). This will be preceded with a single series of 5 consecutive patients (Part A).
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgery utilizing the Kidney Skinn cooling device (Experimental): All patients in Part A, and those randomized to the Kidney Skinn arm in Part B, will receive transplant surgery in the traditional fashion with the exception that the renal allograft will be placed in the cooling device at the initiation of the vascular anastomosis. Cold saline irrigation flowing through the device will be used to maintain renal hypothermia for the duration for the vascular anastomosis. After the vascular clamps are released, the device will be removed.
  Interventions: Device: Kidney cooling device
- Standard transplant surgery practice (No Intervention): Standard transplant surgery per site practice

INTERVENTIONS:
Device: Kidney cooling device — renal cooling device designed to maintain renal hypothermia at or below 5ºC for 60 minutes.
  Other Names: Kidney Skinn
  Arms: Surgery utilizing the Kidney Skinn cooling device

SUMMARY:
Avoiding warm ischemia time during vascular anastomosis of the renal allograft is important to prevent damage. The investigators are studying a cooling device that may control the temperature of the renal allograft during transplant surgery; attempting to keep temperatures at or below 5°C for at least 60 minutes. If found effective, this could eliminate warm ischemia and potentially prevent damage to transplanted kidneys.

DETAILED DESCRIPTION:
Warm ischemia can damage a renal allograft in many different ways often leading to early failure of the kidney transplant and sometimes even death of the transplant recipient. For this reason every effort is made to keep the allograft cold during the removal and transportation, and protocols have been developed to ensure this. Although kidneys are kept below 5°C during transportation, they re-warm rapidly during the transplant surgery. On average, kidneys are exposed to 40 or more minutes of dangerously warm temperatures during transplant surgery.

To avoid damage, it is important to reduce the amount of time it is exposed to warm temperatures. Currently, there are no devices or standardized protocols available to ensure a kidney stays cold during the transplant surgery.

The Principal Investigator has developed Kidney Skinn, a device that may control the temperature of the renal allograft during transplant surgery; keeping allograft temperatures at or below 5°C for at least 60 minutes. If found effective, this could eliminate warm ischemia and potentially prevent damage to transplanted kidneys. The device may also potentially provide retraction and support for the kidney during the transplant operation, making the surgery easier to perform. Additionally, the device may be found to be easily removed once the transplant is complete.

A previous study was conducted with the Kidney Skinn in animals; the next step is to investigate whether the device can perform in the human clinical setting. This study will be done in 2 steps. Part A: a series of consecutive consenting patients to determine device initial safety, and Part B: a single-centre randomized-controlled pilot study of kidney transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age at time of transplant
2. Slated to receive a single cadaveric organ
3. Donor declared by traditional neurological determination of death (NDD)
4. Standard criteria donor (SCD) or Extended criteria donor (ECD)
5. Consent obtained prior to the transplant operation

Exclusion Criteria:

1. Living donor (LD)
2. Donor after cardiocirculatory death (DCD)
3. Highly sensitized patients (those with Panel-reactive antibody or PRA >80%)
4. Recipient of a previous kidney transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Part A: Device design is deemed suitable to move into the traditional feasibility stage (Part B of protocol) | 6 months
  The Kidney Skinn cooling device can be utilized during vascular anastomosis, and the ability of the device to maintain surface and core temperatures of transplant kidneys at <5ºC for the duration of the vascular anastomosis.
Part B: To determine the feasibility of a trial using the Kidney Skinn cooling device to usual care to ameliorate warm ischemia time during kidney transplantation | 2 years
  Feasibility Outcomes will include the following:
  1. Ability to randomize >60% of eligible patients
  2. >75% of patients randomized to the Kidney Skinn arm use the device
  3. 70% of patients randomized to the device (Kidney Skinn) achieve a renal allograft surface temperature of <5C for the duration of the vascular anastomosis.

SECONDARY OUTCOMES:
Proportion of patients who develop delayed graft function (need for dialysis in the first week after transplantation) compared with usual care | 7 days
  Delayed Graft function as defined by the need for dialysis in the first 7 post operative days
Difference in ischemia-reperfusion injury biomarker levels between the intervention and control groups | 7 days
  Urine and serum biomarkers for ischemia-reperfusion injury will be collected at specific key time points pre and post transplantation on all Part B trial participants. Specifically, urine and serum samples for unique markers of kidney injury (KIM-1 & NGAL), inflammation (TNFR1, MCP-1) and fibrosis (suPAR, YKL 40).
Serum creatinine level at discharge from initial hospitalization for transplantation | 5-7 days
  Local laboratory serum creatinine drawn per standard of care on all renal transplant recipients on day of discharge
Differences in achieved renal allograft surface temperature comparing the Kidney Skinn (intervention arm) versus usual care (control arm) | 60 minutes
  For each surgery, K-type 30 gauge thermocouples (each less than 0.25mm in external diameter) will be used in the renal allograft at a depth of 5 mm and 15 mm. This will be to measure surface (cortical) and core (medullary) temperatures, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Skinner, Principal Investigator — Nova Scotia Health Authority; Karthik Tennankore, Principal Investigator — Nova Scotia Health Authority
Locations (1):
- Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No
This is a pilot study